CLINICAL TRIAL: NCT04169490
Title: "A Prospective, Randomized, Double-blind, Placebo Controlled and Comparative Clinical Study Evaluating Scar-management Modalities for Simple and Effective Management of Hyperproliferative (Hypertrophic) Scars and Keloids"
Brief Title: "A Clinical Study Investigating the Effectiveness of OTC Scar-management Modalities"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Center for Clinical and Cosmetic Research (Other)
Collaborators: BirchBioMed Inc. (Unknown)
Responsible Party: Principal Investigator, Mark Steven Nestor, M.D., Ph.D., Director, The Center for Clinical and Cosmetic Research
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCCR 02-2019
Record Dates: First submitted 2019-11-15; First posted 2019-11-20 (Actual); Last update posted 2022-03-21 (Actual); Status verified 2022-03

CONDITIONS: Scar; Keloid; Hypertrophic Scar; Cicatrix
Keywords: Scar; Keloid; Hypertrophic Scar; Cicatrix
MeSH Terms: conditions — Cicatrix; Keloid; Cicatrix, Hypertrophic

STUDY DESIGN:
Intervention Model Description: The study consists of five Treatments across two study Arms of which include a placebo, a 510(k) market-approved "Active" comparator with and without FS2, and two cosmetic, moisturizer formulation variants that have not demonstrated therapeutic efficacy, but are hypothesized to improve the appearance of scar-prone wounds once healed. The Placebo moisturizer serves as the negative control, whereas the silicone gel serves both purposes as a negative control for the FS2 incorporated silicone gel and active comparator for both FS2 silicone gel and the moisturizing products.
Who Masked: Participant, Investigator
Masking Description: This is a double-blinded study, which means that neither the evaluating physician nor the subject will know which treatment is administered. A separate study staff member will administer the treatment, as well as answer questions and discuss any problems prior to starting, and for the duration of, the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- FS2 Emulsion Moisturizer (Experimental): The FS2 Emulsion Moisturizer Arm is comprised of three (3) topical treatments including: Placebo Cream Base Emulsion Moisturizer, FS2 Emulsion Moisturizer and Active Comparator Onion Skin Extract Gel (Mederma). The topical treatments are applied b.d. for 120 days.
  Interventions: Other: Placebo Cream Base Emulsion Moisturizer; Other: FS2 Emulsion Moisturizer; Other: Active Comparator Onion Skin Extract Gel (Mederma)
- Active Comparator + FS2 Emulsion Moisturizer (Experimental): The Active Comparator + FS2 Emulsion Moisturizer Arm is comprised of two (2) topical treatments including: Active Comparator Silicone Gel (Kelo-Cote), and Active Comparator Silicone Gel (Kelo-Cote) + FS2 Emulsion Moisturizer. The topical treatments are applied b.d. for 120 days.
  Interventions: Other: Active Comparator Silicone Gel (Kelo-Cote); Other: Active Comparator Silicone Gel (Kelo-Cote) + FS2 Emulsion Moisturizer

INTERVENTIONS:
Other: Placebo Cream Base Emulsion Moisturizer — Topical placebo white, oil/water emulsion moisturizer applied b.d. for 120 days
  Arms: FS2 Emulsion Moisturizer
Other: FS2 Emulsion Moisturizer — Topical FS2 white, oil/water emulsion moisturizer applied b.d. for 120 days
  Arms: FS2 Emulsion Moisturizer
Other: Active Comparator Onion Skin Extract Gel (Mederma) — Topical onion skin extract gel (Mederma) applied b.d. for 120 days
  Arms: FS2 Emulsion Moisturizer
Other: Active Comparator Silicone Gel (Kelo-Cote) — Topical silicone gel (Kelo-Cote) applied b.d. for 120 days
  Arms: Active Comparator + FS2 Emulsion Moisturizer
Other: Active Comparator Silicone Gel (Kelo-Cote) + FS2 Emulsion Moisturizer — Topical silicone gel (Kelo-Cote) + Topical FS2 white, oil/water emulsion moisturizer applied b.d. for 120 days
  Arms: Active Comparator + FS2 Emulsion Moisturizer

SUMMARY:
A Phase II prospective, randomized, double-blind, placebo controlled and comparative clinical study evaluating hydrogel scar-management modalities for effective management of hyperproliferative scars and keloids.

This is a double-blinded study, which means that neither the evaluating physician nor the subject will know which treatment is administered.

Group selection and assignment will be made at random, with a 2 in 5 chance of receiving a market-approved therapy, and 1 in 5 chance of receiving the placebo. Subjects assigned the placebo-moisturizer will receive a standard hypoallergenic dermatological hydrating cream base. Subjects assigned the silicone gel, will receive a commercially available, active comparator.

DETAILED DESCRIPTION:
A Phase II prospective, randomized, double-blind, placebo controlled and comparative clinical study evaluating hydrogel scar-management modalities for effective management of hyperproliferative scars and keloids. Unlike raised and, or hyperproliferative scars that result from aberrant wound healing, keloids are the result of inherited genetic mutations in a variety of proteins essential to orchestrated wound repair. Whereas hyperproliferative scars may have shared similar abnormalities throughout the repair of a primary injury, they are not predictors of subsequent scarring following scar revision. Keloids on the other hand will return upon excision, and in some cases larger in size than the excised scar tissue. Current treatment options for keloids as well as hypertrophic scars include intralesional corticosteroids, silicone gel sheeting, compression, surgery and adjuvants to surgery, including radiation and cryotherapy.

Onion skin extract, silicone, and a variety of over-the-counter selfcare product options are available for patients with keloids and hypertrophic scars. Despite market approval, robust efficacy data to substantiate product claims is scarce. At best, comparative studies have been able to demonstrate significance between modalities/products. With only a limited number of investigator initiated studies with scar-patients the advancement in this niche, yet expansive, medical sector has been incremental across decades of research. This study is being undertaken to investigate the efficacy and safety of a FS2- moisturizer, and two market-approved scar topical therapies. The FS2- moisturizer is claimed to be substantially equivalent or superior to market approved Onion skin extract (Mederma), and silicone gel (Kelo-Cote)intended to manage and improve hyperproliferative closed scars. The study builds upon a recent study that investigated safety and efficacy of a petrolatum lotion vs. onion-extract gel vs. placebo in subjects with hypertrophic scars and keloids. There two (2) Study Arms and five (5) Treatment Groups. Treatment Groups consist of: placebo moisturizer cream base, Onion skin extract (Mederma), FS2-moisturizer formulations, silicone gel (Kelo-Cote), and an FS2-silicone gel.

This is a double-blinded study, which means that neither the evaluating physician nor the subject will know which treatment is administered. A separate study team member will administer the treatment, as well as answer questions and discuss any problems prior to starting, and for the duration of, the study.

Subjects will be assigned a Treatment Group from those listed above. Group selection and assignment will be made at random, with a 2 in 5 chance of receiving a market-approved therapy, and 1 in 5 chance of receiving the placebo. Subjects assigned the placebo-moisturizer will receive a standard hypoallergenic dermatological hydrating cream base. Subjects assigned the silicone gel, will receive a commercially available, active comparator.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female
2. Adult, Senior (>18 years of age)
3. Healthy or medically stable
4. Keloid or hypertrophic scar
5. Willing and able to follow study requirements
6. Etiology and clinical assessment of the scar indicate that it could benefit from the study treatments

Exclusion Criteria:

1. Subjects who are medically unstable
2. Subjects who are expected to be medically unstable for the duration of the study period and an additional 1-month thereafter
3. Pregnant subjects, or those attempting to become pregnant
4. Subjects with known immunosuppression or immunosuppressive illness
5. Subjects with uncontrolled diabetes or autoimmune disorders
6. Subjects with known sensitivity to ingredients in the test-treatment products
7. Subjects who are enrolled in another scar study and/or plan to receive or are receiving scar treatments other than study treatment during the trial period
8. Subjects who have received scar treatment, including any investigational treatment, within one month of the first day of study treatment
9. Subjects with any skin conditions or taking any medications that may interfere with the study medication
10. Subjects who had any clinical evidence of severe ongoing or prolonged depression, mental illness, and/or who has demonstrated evidence of drug abuse
11. Any other diagnosis, condition, physical or geographical limitation that may render, or increases the likelihood of rendering, the Subject unable to complete the entire study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-02-07 (Actual); Primary Completion 2020-09-04 (Actual); Study Completion 2020-11-03 (Actual)

PRIMARY OUTCOMES:
Vancouver Scar Scale (VSS) | 180 Days
  Investigator assessment of target scar or keloid using the Vancouver Scar Scale (VSS). Scale parameters include: Pigmentation (0-2), Vascularity (0-3), Pliability (0-5), and Height (0-3). Scale measurements include: minimum score of 0 = normal to a maximum score of 2, 3 or 5 depending on the parameter measured.
Patient and Observer Scar Assessment Scale (POSAS) | 180 Days
  Investigator assessment of target scar or keloid using the Patient and Observer Scar Assessment Scale (POSAS). Scale parameters include: Vascularity, Pigmentation, Thickness, Relief, Pliability, and Surface Area. Scale measurements include: minimum score of 1 = normal skin to a maximum score of 10 = worst scar imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nestor, M.D., Ph.D., Principal Investigator — The Center for Clinical and Cosmetic Research
Locations (1):
- The Center for Clinical and Cosmetic Research, Aventura, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: BirchBioMed Inc. — http://www.birchbiomed.com
- See also: Mederma — https://www.mederma.com/
- See also: Kelo-Cote — https://kelocote.com/